CLINICAL TRIAL: NCT04735276
Title: MRI Study of the Gastric Insufflation After High-flow Nasal Oxygen (HFNO)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Benjamin Javillier, Principal Investigator, University of Liege
Other Study IDs: Optirm
Record Dates: First submitted 2021-01-25; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: HFNO for 5 min — 1st basic MRI then HFNO for 5 min with mouth closed breathing and 2nd MRI. Analysis of the surface of the gastric antrum.

SUMMARY:
HFNO CAN BE USED AS A PREOXYGENATION TECHNIQUE BUT IS IT A SAFE TECHNIQUE IN TERMS OF GASTRIC INSUFFLATION?

DETAILED DESCRIPTION:
The objective of this study is to evaluate by MRI whether the stomach is insufflated during HFNO use in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Adults Volunteers

Exclusion Criteria:

* Pregnancy
* Claustrophobia
* Gastric surgery
* Gastric pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adult volunteers
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of the antero-posterior and cranio-caudal diameters of the gastric antrum | through study completion, an average of 1 year
  surface of the gastric antrum